CLINICAL TRIAL: NCT04735445
Title: IMPACt of an Enhanced Screening Program on the Detection of Non-AIDS NEOplasms in Patients With Human Immunodeficiency Virus (HIV) Infection
Brief Title: IMPACt of an Enhanced Screening Program on the Detection of Non-AIDS NEOplasms in HIV Patients
Acronym: IMPACNEO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Felix Gutierrez (Other)
Collaborators: Instituto de Salud Carlos III (Other Government); Hospital General Universitario Reina Sofía de Murcia (Other); Hospital Universitario Reina Sofia de Cordoba (Other Government); Hospital General Universitario de Alicante (Other); Hospital Clinic of Barcelona (Other); Hospital Universitario Ramon y Cajal (Other); Hospital General Universitario Santa Lucia (Other); Fundación de Investigación Biomédica - Hospital Universitario de La Princesa (Other); Hospital Universitario de Guadalajara (Unknown); Hospital Universitario Virgen de la Arrixaca (Other); Parc Taulí Hospital Universitari (Other); Hospital Universitario La Fe (Other); Germans Trias i Pujol Hospital (Other); Complejo Hospitalario Universitario de Albacete (Other); Hospital Universitario Fundación Alcorcón (Other); Hospital General Universitario Elche (Other)
Responsible Party: Sponsor-Investigator, Felix Gutierrez, Principal Investigator, Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana
Organization: Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: IMPACNEO
Record Dates: First submitted 2021-01-27; First posted 2021-02-03 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-02

CONDITIONS: HIV/AIDS; Cancer
Keywords: HIV; Neoplasm; Screening; Early diagnosis
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Neoplasms; Disease | interventions — Biopsy; Mammography; Occult Blood; Tomography, X-Ray Computed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional screening (Active Comparator): Standard screening in the participating centers, adjusted to the recommendations of the European AIDS Society (EACS).
  Interventions: Diagnostic Test: Digital rectal exam and / or anal cytology (day 1 and after 36 months); Diagnostic Test: Cervical cytology and cervical sample for HPV detection (day 1 and after 36 months); Diagnostic Test: Appointment for mammography (day 1 and after 36 months); Diagnostic Test: Semestral appointment for liver ultrasound; Diagnostic Test: Fecal occult blood test (day 1 and after 36 months); Diagnostic Test: Digital rectal exam and PSA determination (day 1 and after 36 months)
- Enhanced screening (Experimental): Expanded screening for early detection of lung, liver, anal, cervical, breast, prostate, colorectal and skin cancer.
  Interventions: Diagnostic Test: Semestral digital rectal exam and / or anal cytology if abnormal → ANOSCOPY with biopsy; Diagnostic Test: Semestral cervical cytology and cervical sample for HPV detection; Diagnostic Test: Annual appointment for mammography; Diagnostic Test: Semestral appointment for liver ultrasound; Diagnostic Test: Semestral blood collection for alpha-fetoprotein and others hepatic biomarkers determination; Diagnostic Test: Annual fecal occult blood test; Diagnostic Test: Annual digital rectal exam and PSA determination; Diagnostic Test: Annual appointment for low dose computed tomography for lung screening; Diagnostic Test: Annual general inspection for skin lesions suggestive of malignancy

INTERVENTIONS:
Diagnostic Test: Digital rectal exam and / or anal cytology (day 1 and after 36 months) — For anal screening in MSM man or woman with abnormal cervical cytology, genital warts or having anal sex (day 1 and after 36 months)
  Arms: Conventional screening
Diagnostic Test: Semestral digital rectal exam and / or anal cytology if abnormal → ANOSCOPY with biopsy — For anal screening in MSM man or woman with abnormal cervical cytology, genital warts or having anal sex (semestral)
  Arms: Enhanced screening
Diagnostic Test: Cervical cytology and cervical sample for HPV detection (day 1 and after 36 months) — For Cervix Screening in sexually active woman (day 1 and after 36 months)
  Arms: Conventional screening
Diagnostic Test: Semestral cervical cytology and cervical sample for HPV detection — For Cervix Screening in sexually active woman (semestral)
  Arms: Enhanced screening
Diagnostic Test: Appointment for mammography (day 1 and after 36 months) — For Breast Screening in woman between 50-70 years old (day 1 and after 36 months)
  Arms: Conventional screening
Diagnostic Test: Annual appointment for mammography — For Breast Screening in woman between 45-70 years old (annual)
  Arms: Enhanced screening
Diagnostic Test: Semestral appointment for liver ultrasound — For Hepatic Screening:
  Cirrhosis or Chronic HBV, and meet any of the following risk factors:
  * Asian male> 40 years old
  * Asian woman> 50 years old
  * African man or woman
  * HCC family history
  Arms: Conventional screening
Diagnostic Test: Semestral appointment for liver ultrasound — Having chronic liver disease with fibrosis ≥ F3 or Presents chronic HBV
  Arms: Enhanced screening
Diagnostic Test: Semestral blood collection for alpha-fetoprotein and others hepatic biomarkers determination — Having chronic liver disease with fibrosis ≥ F3 or Presents chronic HBV
  Arms: Enhanced screening
Diagnostic Test: Fecal occult blood test (day 1 and after 36 months) — For Colon Screening:
  Age between 50-70 years old
  Arms: Conventional screening
Diagnostic Test: Annual fecal occult blood test — For Colon Screening:
  Age older than 40 years
  Arms: Enhanced screening
Diagnostic Test: Digital rectal exam and PSA determination (day 1 and after 36 months) — For Prostate Screening:
  Man older than 50 years
  Arms: Conventional screening
Diagnostic Test: Annual digital rectal exam and PSA determination — For Prostate Screening:
  Man older than 50 years
  Arms: Enhanced screening
Diagnostic Test: Annual appointment for low dose computed tomography for lung screening — For Lung Screening: should accomplish
  ALL the following criteria:
  * Age > 40 years
  * Active smoker or former smoker<3 years, with IPY ≥20. IPY: index of packages-year: nº packages that smoke per day x nº years smoking
  * No contraindications for thoracic surgery
  * No lung infection in the last 2 months
  Arms: Enhanced screening
Diagnostic Test: Annual general inspection for skin lesions suggestive of malignancy — For Skin Screening:
  Woman ≥18 years Man ≥40 years
  Arms: Enhanced screening

SUMMARY:
Introduction: The incidence of malignancies is higher in the HIV-infected population than in the general population, and it is already one of the leading causes of death in people living with the virus. It is estimated that the situation will be aggravated by the progressive aging of the HIV-infected population. Early diagnosis through enhanced cancer screening can be critical in reducing mortality, but may increase expenditure and harms associated with adverse events. This strategy should then be considered only when the benefits clearly outweigh the harms. There are currently no studies on expanded cancer screening in patients with HIV, and available information from the point of view of costeffectiveness or cost-utility is scarce.

Hypothesis: An enhanced program for non-aids cancer screening in patients with HIV can lead to early diagnosis and improve the prognosis of these patients, with an acceptable rate of unnecessary interventions and being cost-effective.

Objectives: To evaluate the efficacy, safety and efficiency of an enhanced screening program for the early diagnosis of cancer in HIV patients compared to standard practice within the cohort of the National AIDS Research Network (CoRIS).

Specific objectives: 1) To compare the incidence of early diagnosed cancer with enhanced screening versus conventional screening; 2) To assess the incidence of early diagnosed cancer and its overall incidence in the CoRIS cohort; 3) To analyze safety of the program: adverse events and unnecessary interventions; 4) To compare the obtained data stratifying by gender and 5) To analyze the cost-utility of the program.

Expected results: 1) To generate scientific evidence to inform decision makers on the advisability of implementing an enhanced screening program of cancer in HIV-infected patients; 2) To broaden knowledge about the programs of early detection of cancer in vulnerable populations and their economic evaluation from the perspective of the National Health Service.

DETAILED DESCRIPTION:
Non-AIDS-Defining Cancers (NADCs) are an important cause of morbidity and mortality in the population living with the human immunodeficiency virus (PLHIV), being currently one of the most frequent causes of death. Due to several reasons, the incidence of this type of tumors in PLHIV has increased 2-3 times with respect to the general population (GP). In a recent systematic review, with more than 600,000 PLHIV and 10,891 new cases of cancer, it is demonstrated how the incidence of NADCs has progressively increased since the introduction of combined antiretroviral therapy (ART), probably reflecting better viral-immune control and aging associated with the increase in overall survival of patients living with the virus. The most frequent cancers are lung cancer, hepatocellular carcinoma, anal carcinoma and cervical carcinoma, although some studies have suggested that there could also be a higher incidence and / or severity of other malignant tumors, such as breast cancer, prostate, colorectal or skin, including melanomas. In the era of ART, lung cancer has become the most frequent and deadliest cause of non-AIDS-associated cancer in PLHIV, and greater lethality has been documented in PLHIV than in GP.

The causes of this increased incidence of NADCs are not well known and there are several factors that could influence, including the oncogenic effects of the virus, immunosuppression, chronic inflammation and immune activation, ART exposure, higher rates of coinfection with other oncogenic viruses and traditional cancer risk factors such as smoking. It is estimated that at least 1 in 3 PLHIV will die due to malignant neoplasms in the coming years. There is currently no consensus on the best screening strategies in this population, strategies that seem increasingly necessary considering the progressive aging of the infected population and the increase in the incidence of these neoplasms.

In some of the clinical practice guidelines in PLHIV, such as the Spanish Gesida or other European ones, the screening strategies for neoplasms recommended in GP have been incorporated, in which they have shown benefit in terms of mortality or greater probabilities of therapeutic success. However, these benefits have not been confirmed in PLHIV, in which this type of strategy could be insufficient.

Moreover, there are currently no established recommendations for GP screening on two of the main neoplasms of PLHIV, such as lung and anal. For this reason, it is necessary to generate scientific evidence that determines which is the most convenient strategy to reduce the morbidity and mortality associated with NADCs in PLHIV. Then, the evaluation of an enhanced program of screening by conducting a clinical trial, in which patients are randomized to one of the two strategies (enhanced screening versus standard of care practice), is the ideal design to generate scientific evidence. This knowledge could be useful to determine if the benefits of the enhanced screening outweighs the harms and if it is cost-effective for the National Health Service.

Objectives:

General objectives: To evaluate the efficacy, safety and efficiency of an expanded screening program for the early diagnosis of cancer in patients with HIV compared to usual practice, within the framework of the Spanish AIDS Research Network (RIS).

Specific objectives: 1) To compare the incidence of early diagnosed cancer with extended screening versus usual practice; 2) To estimate the incidence of early diagnosed cancer and its overall incidence in the CoRIS cohort; 3) To analyze safety of the program: adverse events and unnecessary interventions; 4) To compare the incidence data described above stratifying by gender and 5) To analyze the cost-utility of the extended screening.

Early detection of cancer would entail clinical benefits, both in terms of survival and quality of life, for the population with HIV. The evaluation of the cost-utility of the program is also a main objective, since the benefits of therapy for cancer in the earliest stages should compensate for the use of the additional resources of the National Health System.

Methodology: Research project that includes randomization by patient, stratified according to sex, to one of the following groups:

1. Enhanced intervention group: expanded screening for early detection of lung, liver, anal, cervical, breast, prostate, colorectal and skin cancer.
2. Conventional intervention group: standard screening in the participating centers, adjusted to the recommendations of the European AIDS Society (EACS).

Work plan and timeline

This project is based on a collaborative methodology in which all groups work in a coordinated manner, under the direction of the Principal Investigator, Dr. Félix Gutiérrez. The tasks that make up this project are broken down below:

1. Recruitment of patients and randomization according to the sex of each patient to a conventional intervention or an extended intervention. This phase is already started in some of the centers that make up the consortium, but it must continue to reach the desired sample size. Depending on whether the patients are assigned to the conventional screening group or the extended screening group, their inclusion in the following tasks will be different.
2. Completion of the questionnaires (annual) on sociodemographic and toxic data in each of the participating centers.
3. Blood samples withdrawal and storage of plasma for ulterior determination of biomarkers annually.
4. The digital examination and anal (semi-annual) cytology, cervical cytology (semi-annual) will be performed in the HIV Units of the participating centers.
5. The General Inspection in search of skin lesions suggestive of malignancy on an annual basis will be carried out in the HIV Units of the participating centers that will be previously trained for it. In case of suspicion, it will be referred to the specialist of each center.
6. The semi-annual monitoring of the clinical trial will be carried out by the CRO contracted for that purpose.
7. At 30 months, the telematic session for closing the trial will be held.
8. Statistical analysis of the data. The analysis of the data will be carried out transversely after the first year, after the second and after the third year, where the final conclusions of the study can be established.
9. Dissemination of the results during the last 3 months: communications to congresses and writing of articles. Proposal for inclusion in Clinical Guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Male ≥40 years or woman ≥18 years
* Informed Consent signed

Exclusion Criteria:

* Active AIDS defining disease
* Antecedent of cancer
* Terminal disease
* Pregnancy or breastfeeding
* Patient rejection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Both genders should be represented in a real incidence estimation of Spanish population.
Enrollment: 4638 (Estimated)
Dates: Start 2019-11-11 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Non-AIDS defining cancers incidence | through study completion, an average of 1 year
  The incidence of different neoplasms not considered as AIDS defining cancers compared between two arms
Survival rate | through study completion, an average of 1 year
  Comparison in survival terms between conventional and enhanced screening arms

SECONDARY OUTCOMES:
Safety of the screening: adverse events | through study completion, an average of 1 year
  Analyze the safety of the screening program, analyzing its adverse events, including those unnecessary interventions
Cost-efectiveness | through study completion, an average of 1 year
  Analyze the cost-utility ratio of the extended screening program.

CONTACTS AND LOCATIONS:
Overall Officials: Félix Gutiérrez-Rodero, PhD, Principal Investigator — Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana
Locations (1):
- Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana, Elche, Alicante, Spain

REFERENCES:
- [Result] Lopez C, Masia M, Padilla S, Aquilino A, Bas C, Gutierrez F. [Deaths due to non-AIDS diseases among HIV infected patients: A 14-year study (1998-2011)]. Enferm Infecc Microbiol Clin. 2016 Apr;34(4):222-7. doi: 10.1016/j.eimc.2015.04.010. Epub 2015 Jun 18. Spanish. PMID 26093959
- [Result] Garcia-Abellan J, Del Rio L, Garcia JA, Padilla S, Vivancos MJ, Del Romero J, Asensi V, Hernando A, Garcia-Fraile L, Masia M, Gutierrez F; la Cohorte de la Red Nacional de Sida (CoRIS). Risk of cancer in HIV-infected patients in Spain, 2004-2015. The CoRIS cohort study. Enferm Infecc Microbiol Clin (Engl Ed). 2019 Oct;37(8):502-508. doi: 10.1016/j.eimc.2018.11.011. Epub 2019 Jan 22. English, Spanish. PMID 30679001
- [Result] Smith CJ, Ryom L, Weber R, Morlat P, Pradier C, Reiss P, Kowalska JD, de Wit S, Law M, el Sadr W, Kirk O, Friis-Moller N, Monforte Ad, Phillips AN, Sabin CA, Lundgren JD; D:A:D Study Group. Trends in underlying causes of death in people with HIV from 1999 to 2011 (D:A:D): a multicohort collaboration. Lancet. 2014 Jul 19;384(9939):241-8. doi: 10.1016/S0140-6736(14)60604-8. PMID 25042234
- [Result] Shiels MS, Cole SR, Kirk GD, Poole C. A meta-analysis of the incidence of non-AIDS cancers in HIV-infected individuals. J Acquir Immune Defic Syndr. 2009 Dec;52(5):611-22. doi: 10.1097/QAI.0b013e3181b327ca. PMID 19770804
- [Result] Grulich AE, van Leeuwen MT, Falster MO, Vajdic CM. Incidence of cancers in people with HIV/AIDS compared with immunosuppressed transplant recipients: a meta-analysis. Lancet. 2007 Jul 7;370(9581):59-67. doi: 10.1016/S0140-6736(07)61050-2. PMID 17617273
- [Result] Althoff KN, McGinnis KA, Wyatt CM, Freiberg MS, Gilbert C, Oursler KK, Rimland D, Rodriguez-Barradas MC, Dubrow R, Park LS, Skanderson M, Shiels MS, Gange SJ, Gebo KA, Justice AC; Veterans Aging Cohort Study (VACS). Comparison of risk and age at diagnosis of myocardial infarction, end-stage renal disease, and non-AIDS-defining cancer in HIV-infected versus uninfected adults. Clin Infect Dis. 2015 Feb 15;60(4):627-38. doi: 10.1093/cid/ciu869. Epub 2014 Oct 30. PMID 25362204
- [Result] Cobucci RN, Lima PH, de Souza PC, Costa VV, Cornetta Mda C, Fernandes JV, Goncalves AK. Assessing the impact of HAART on the incidence of defining and non-defining AIDS cancers among patients with HIV/AIDS: a systematic review. J Infect Public Health. 2015 Jan-Feb;8(1):1-10. doi: 10.1016/j.jiph.2014.08.003. Epub 2014 Oct 5. PMID 25294086
- [Result] Masia M, Padilla S, Alvarez D, Lopez JC, Santos I, Soriano V, Hernandez-Quero J, Santos J, Tural C, del Amo J, Gutierrez F; CoRIS. Risk, predictors, and mortality associated with non-AIDS events in newly diagnosed HIV-infected patients: role of antiretroviral therapy. AIDS. 2013 Jan 14;27(2):181-9. doi: 10.1097/QAD.0b013e32835a1156. PMID 23018442
- [Result] Patel P, Hanson DL, Sullivan PS, Novak RM, Moorman AC, Tong TC, Holmberg SD, Brooks JT; Adult and Adolescent Spectrum of Disease Project and HIV Outpatient Study Investigators. Incidence of types of cancer among HIV-infected persons compared with the general population in the United States, 1992-2003. Ann Intern Med. 2008 May 20;148(10):728-36. doi: 10.7326/0003-4819-148-10-200805200-00005. PMID 18490686
- [Result] Shiels MS, Engels EA. Evolving epidemiology of HIV-associated malignancies. Curr Opin HIV AIDS. 2017 Jan;12(1):6-11. doi: 10.1097/COH.0000000000000327. PMID 27749369
- [Result] Croxford S, Kitching A, Desai S, Kall M, Edelstein M, Skingsley A, Burns F, Copas A, Brown AE, Sullivan AK, Delpech V. Mortality and causes of death in people diagnosed with HIV in the era of highly active antiretroviral therapy compared with the general population: an analysis of a national observational cohort. Lancet Public Health. 2017 Jan;2(1):e35-e46. doi: 10.1016/S2468-2667(16)30020-2. Epub 2016 Dec 15. PMID 29249478
- [Result] Wang YH, Shen XD. Human immunodeficiency virus infection and mortality risk among lung cancer patients: A systematic review and meta-analysis. Medicine (Baltimore). 2018 Apr;97(15):e0361. doi: 10.1097/MD.0000000000010361. PMID 29642182
- [Result] Trickey A, May MT, Gill MJ, Grabar S, Vehreschild J, Wit FWNM, Bonnet F, Cavassini M, Abgrall S, Berenguer J, Wyen C, Reiss P, Grabmeier-Pfistershammer K, Guest JL, Shepherd L, Teira R, d'Arminio Monforte A, Del Amo J, Justice A, Costagliola D, Sterne JAC. Cause-specific mortality after diagnosis of cancer among HIV-positive patients: A collaborative analysis of cohort studies. Int J Cancer. 2020 Jun 1;146(11):3134-3146. doi: 10.1002/ijc.32895. Epub 2020 Mar 12. PMID 32003460
- [Result] Santos J, Valencia E; Panel de Expertos de GeSIDA. [Consensus statement on the clinical management of non-AIDS defining malignancies. GeSIDA expert panel]. Enferm Infecc Microbiol Clin. 2014 Oct;32(8):515-22. doi: 10.1016/j.eimc.2014.04.008. Epub 2014 Jun 20. Spanish. PMID 24953385
- [Result] GBD 2015 HIV Collaborators. Estimates of global, regional, and national incidence, prevalence, and mortality of HIV, 1980-2015: the Global Burden of Disease Study 2015. Lancet HIV. 2016 Aug;3(8):e361-e387. doi: 10.1016/S2352-3018(16)30087-X. Epub 2016 Jul 19. PMID 27470028
- [Result] Rubinstein PG, Aboulafia DM, Zloza A. Malignancies in HIV/AIDS: from epidemiology to therapeutic challenges. AIDS. 2014 Feb 20;28(4):453-65. doi: 10.1097/QAD.0000000000000071. PMID 24401642
- [Result] Ryom L, Cotter A, De Miguel R, Beguelin C, Podlekareva D, Arribas JR, Marzolini C, Mallon P, Rauch A, Kirk O, Molina JM, Guaraldi G, Winston A, Bhagani S, Cinque P, Kowalska JD, Collins S, Battegay M; EACS Governing Board. 2019 update of the European AIDS Clinical Society Guidelines for treatment of people living with HIV version 10.0. HIV Med. 2020 Nov;21(10):617-624. doi: 10.1111/hiv.12878. Epub 2020 Sep 3. PMID 32885559
- [Derived] Gutierrez F, Lopez L, Galera C, Tiraboschi JM, Portu J, Garcia-Fraile L, Garcia Del Toro M, Bernal E, Rivero A, Garcia-Abellan J, Flores J, Gonzalez-Cordon A, Martinez O, Bravo J, Rosado D, Montero M, Sirera G, Torralba M, Galindo MJ, Macias J, Gonzalez-Cuello I, Boix V, Vivancos MJ, Dios P, Blanco JR, Padilla S, Fernandez-Gonzalez M, Gutierrez-Ortiz de la Tabla A, Martinez E, Masia M; IMPAC-Neo Study Group. Early Detection of Cancer and Precancerous Lesions in Persons With HIV Through a Comprehensive Cancer Screening Protocol. Clin Infect Dis. 2025 Feb 24;80(2):371-380. doi: 10.1093/cid/ciae359. PMID 38959300
- [Derived] Masia M, Padilla S, Estan G, Portu J, Silva A, Rivero A, Gonzalez-Cordon A, Garcia-Fraile L, Martinez O, Bernal E, Galera C, Boix Martinez V, Macias J, Montero M, Garcia-Rosado D, Vivancos-Gallego MJ, Llenas-Garcia J, Torralba M, Garcia JA, Agullo V, Fernandez-Gonzalez M, Gutierrez F, Martinez E; IMPAC-NEO Study Group. Impact of an enhanced screening program on the detection of non-AIDS neoplasias in patients with human immunodeficiency virus infection. Trials. 2021 Nov 27;22(1):851. doi: 10.1186/s13063-021-05777-6. PMID 34838115